CLINICAL TRIAL: NCT05943262
Title: Record Voxel Rate Nonlinear Optical Microscope to Unravel Brain Connectome and Signaling
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202302070RIND
Record Dates: First submitted 2023-06-18; First posted 2023-07-13 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-05

CONDITIONS: Brain Tumor; Brain Cancer
Keywords: brain tumor; brain cancer
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- mesoscale nonlinear optical microscope + whole-mount H&E & IHC staining protocol
  Interventions: Device: mesoscale nonlinear optical microscope

INTERVENTIONS:
Device: mesoscale nonlinear optical microscope — The mesoscale nonlinear optical microscope based on the principles of nonlinear optics and computed-algorithms can acquire large-area image within few minutes.

SUMMARY:
The research aims to develop a novel pathological technology, including rapid whole-mount tissue H&E & IHC staining protocol and high-resolution nonlinear optical microscopy imaging system, to intraoperatively assess brain tumor grade, types and other biological parameters.

DETAILED DESCRIPTION:
Brain tumors, especially like glioma, the infiltrative growth pattern resulted in an indistinct margin against normal brain tissues. Surgery is currently the most effective method in prolonging patient's survival, the extent of tumor resection is therefore crucial to the overall outcome. Distinguishing the tumor type and grading can help neurosurgeons plan the intraoperative surgical strategies to cure the suffered patients. Feasible solutions to improve the extent of resections including fluorescence-guided surgery and intraoperative MR imaging are relatively indirect to judge the completeness of tumor resection and its margin; considering means like Moh's surgery performed in the dermatological practice, though it is reasonable to look at the resection proportion by pathological interpretation, it is very time consuming. Besides, many kinds of brain tumors can't be classified only by the outcomes of frozen pathology. There are several related studies trying to solve the problem, but the judgment criteria is not sufficient to meet the standard of modern pathological diagnosis. The research aims to acquire images by optical microscopy from both H&E and IHC stained tissues, and to compare those images with slides obtained by standard pathological workflow in order to achieve accurate and rapid assessment of tumor categories and grading.

ELIGIBILITY:
Inclusion Criteria:

1. Patients older than the age of 20 with diagnosis of brain tumor (both newly-diagnosed or recurrent) who are suitable and willing to receive resection surgery.

Exclusion Criteria:

1. Patients who cannot give consent to participate in the study.
2. The tumor samples failed to give a conclusive pathological diagnosis by standard pathological workflow.
3. Patients who only receives biopsy surgery rather than resection surgery.
4. Significant post-irradiation effect or radiation necrosis reported in the pathological examination.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients older than the age of 20 with diagnosis of brain tumor (both newly-diagnosed or recurrent) who are suitable and willing to receive resection surgery will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Develop a standard whole-mount tissue processing protocol | 3 years
  In this research, the investigators will try to create a standard staining protocol to perform rapid whole-mount H&E and IHC staining on surgical brain tumor specimens, so that the cell morphology (ex: cell shape, cell size, etc) and cell types (ex: astrocytes, oligodendrocytes, T-cells, B-cells, etc) in the images of those tissues can be observed via nonlinear optical microscopy, and the treatment strategy can be set based on subtyping and grading the brain tumors by the pathologists.
Obtain images from H&E and IHC stained brain tumor tissues by nonlinear optical microscopy | 3 years
  Images of brain tumor specimens will be taken by nonlinear optical microscopy and a image database of brain tumors can be created (ex: cell shape, cell size and cell density of different cells in human brain tissues).

SECONDARY OUTCOMES:
Distinguish between normal tissue and brain tumor and determine the extent and grade of the brain tumors | 3 years
  By interpreting the images acquired from nonlinear optical microscope of the two staining methods and the images obtained by bright field microscope for pathologists with standard procedures, an attempt is made to distinguish between normal tissue and brain tumor and determine the extent and grade of those brain tumors (depending on tumor characteristics, such as hypercellularity, microvascular proliferation, necrosis, etc).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Surgery, National Taiwan University Hospital and College of Medicine, National Taiwan University, Taipei, Taiwan